CLINICAL TRIAL: NCT03394612
Title: A Phase II, Prospective, Intra-patient Randomised Controlled, Multicentre Study to Evaluate the Safety and Efficacy of an Autologous Bio-engineered Dermo-epidermal Skin Substitute (EHSG-KF) for the Treatment of Full-Thickness Defects in Adults and Children in Comparison to Autologous Split-thickness Skin Grafts (STSG)
Brief Title: Study With an Autologous Dermo-epidermal Skin Substitute for the Treatment of Full-Thickness Skin Defects in Adults and Children
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CUTISS AG (Industry)
Collaborators: Wyss Zurich (Unknown); Julius Clinical (Industry); Sintesi Research Srl (Industry); University Hospital, Zürich (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBRU-dS-RAC-PII
Record Dates: First submitted 2017-12-07; First posted 2018-01-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-12

CONDITIONS: Skin Wound
Keywords: Scar; Skin; Wound Healing; Tissue Engineering; Dermis; Epidermis
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Option 1 (Other): Location A is the experimental area and Location B is the control area.
  Interventions: Biological: EHSG-KF; Biological: STSG
- Option 2 (Other): Location A is the control area and Location B is the experimental area.
  Interventions: Biological: EHSG-KF; Biological: STSG

INTERVENTIONS:
Biological: EHSG-KF — Transplantation of autologous dermo-epidermal skin substitute EHSG-KF to the experimental area
  Other Names: denovoSkin
Biological: STSG — Transplantation of autologous split-thickness skin graft to the control area
  Other Names: Split-thickness skin graft

SUMMARY:
This phase II trial aims to evaluate the efficacy and safety of EHSG-KF (synonym denovoSkin) in comparison to meshed STSG in adults and children with full-thickness Skin defects.

DETAILED DESCRIPTION:
This multicentre phase II clinical trial will target adults and children with fullt-thickness skin defects to elucidate the benefit of a tissue-engineered autologous skin substitute. Particular emphasis, apart from safety, will be placed on efficacy, e.g. scar quality, in comparison to meshed STSG.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥1 years of age
* Large full-thickness defects that require coverage after excision of: Scars, Benign skin tumors (e.g. neurofibroma), Melanocytic nevus (e.g. giant nevus), Gender reassignment surgery, Soft tissue defect after trauma, Soft tissue defect after infection and debridement (e.g necrotizingn fascitis, hidadentitis suppurativa, purpura fulminans), Flap donorsite (e.g. radial forearm flap)
* Minimal areas requiring coverage (not counting the head and neck area for study patients in The Netherlands): 1-5 years: minimum 9cm2, 6-16 years: minimum 25cm2, >16 years: minimum 45cm2
* Signed Informed consent

Exclusion Criteria:

* Patients tested positive for HBV, HCV, syphilis or HIV
* Patients with known underlying or concomitant medical conditions that may interfere with normal wound healing (e.g. systemic skin and connective tissue diseases, any kind of congenital defect of metabolism including insulin-dependent diabetes mellitus, Cushing syndrome or disease, scurvy, chronic hypothyroidism, congenital or acquired immunosuppressive condition, chronic renal failure, or chronic hepatic dysfunction (Child-Pugh class B or C), severe malnutrition, or other concomitant illness which, in the opinion of the Investigator, has the potential to significantly delay wound healing)
* Severe drug and alcohol abuse
* Pre-existing coagulation disorders as defined by INR outside its normal value, PTT >ULN and fibrinogen <LLN prior to the current hospital admission and / or at the Investigator's discretion
* Patients with known allergies to amphotericin B, gentamicin, penicillin, streptomycin, or bovine collagen
* Previous enrolment of the patient into the current phase II study
* Participation of the patient in another study with conflicting endpoints within 30 days preceding and during the present study
* Patients expected not to comply with the study protocol (including patients with severe cognitive dysfunction/impairment and severe psychiatric disorders)
* Pregnant or breast feeding females
* Intention to become pregnant during the clinical course of the study (12 months)
* Enrolment of the Investigator, his/her family members, employees and other dependent persons

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of EHSG-KF in comparison to STSG based on the assessment of scar quality | 3 months post grafting
  Efficacy of EHSG-KF in comparison to STSG based on the assessment of scar quality, using the POSAS ("Patient and Observer Scar Assessment Scale"). The reported Observer Total Score can range from 1 (best) to 10 (worst).

SECONDARY OUTCOMES:
Efficacy of EHSG-KF in comparison to STSG based on the assessment of scar quality | 3 months and 1 year +/- 30 days post grafting
  Evaluation of scar quality at experimental area and control area, using Cutometer for elasticity measurement
Efficacy of EHSG-KF in comparison to STSG based on the assessment of scar quality | 3 months and 1 year +/- 30 days post grafting
  Evaluation of scar quality at experimental area and control area, using POSAS ("Patient and Observer Scar Assessment Scale") Observer Total Score
Efficacy of EHSG-KF in comparison to STSG based on the assessment of scar quality | 3 months and 1 year +/- 30 days post grafting
  Evaluation of scar quality at experimental area and control area, using POSAS ("Patient and Observer Scar Assessment Scale") Patient Items and Total Score
A Efficacy of EHSG-KF in comparison to STSG based on the assessment of scar quality | 3 months and 1 year +/- 30 days post grafting
  Evaluation of scar quality at experimental area and control area, using Colormeter for skin colour measurement,.
Efficacy of EHSG-KF in comparison to STSG based on the assessment of epithelialisation | 28 +/- 3 days post grafting
  Evaluation of efficacy at experimental area and control area, calculating the epithelialized area as percentage of the total grafted area.
Efficacy of EHSG-KF in comparison to STSG based on the assessment of graft take. | 4-11 days post grafting
  Evaluation of efficacy at experimental area and control area, assessed by the analysis of the graft take
Efficacy of EHSG-KF in comparison to STSG based on the assessment of quality of life. | 1 +/- 30 days year post grafting
  Evaluation of efficacy of experimental and control treatment, assessed by quality of life questionnaires ("Pediatric quality of life inventory")
Efficacy of EHSG-KF in comparison to STSG based on the assessment of quality of life. | 1 +/- 30 days year post grafting
  Evaluation of efficacy of experimental and control treatment, assessed by quality of life questionnaires ("Patient Observer Scar Assessment Scale")
Efficacy of EHSG-KF in comparison to STSG based on the assessment of quality of life. | 1 +/- 30 days year post grafting
  Evaluation of efficacy of experimental and control treatment, assessed by quality of life questionnaires ("EuroQuol 5 dimensions questionnaire")
Efficacy of EHSG-KF in comparison to STSG based on the assessment of quality of life. | 1 +/- 30 days year post grafting
  Evaluation of efficacy of experimental and control treatment, assessed by quality of life questionnaires ("Burn Specific Health Scale Brief")
Safety of EHSG-KF in comparison to STSG based on the assessment of infection rate. | 4-11 days and 19-23 days post grafting
  Evaluation of safety at experimental area and control area based on the infection rate, assessed by using wound swabs and clinical evaluation.
Safety of EHSG-KF in comparison to STSG based on the assessment of adverse events. | through study completion, an average of 3 years
  Evaluation of safety at experimental area and control area, assessed by the type and number of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Sc, Prof., Study Chair — University Children's Hospital, Zurich
Locations (7):
- Italy (3):
  - Chirurgia Plastica e Centro Ustioni Azienda Ospedaliera di Rilievo Nazionale A. Cardarelli, Napoli
  - Unità di Chirurgia Plastica e Ustioni Ospedale Santobono, Napoli
  - U.O.C. Grandi Ustionati Azienda Ospedale Università Padova, Padua
- Netherlands (2):
  - Dept. of Plastic, Reconstructive and Hand Surgery, VU University Medical Center, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
- Switzerland (2):
  - University Children's Hospital Zurich, Zurich
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schiestl C, Neuhaus K, Meuli M, Farkas M, Hartmann-Fritsch F, Elrod J, Bressan J, Reichmann E, Bottcher-Haberzeth S. Long-Term Outcomes of a Cultured Autologous Dermo-Epidermal Skin Substitute in Children: 5-Year Results of a Phase I Clinical Trial. J Burn Care Res. 2025 Mar 4;46(2):326-334. doi: 10.1093/jbcr/irae150. PMID 39115183